CLINICAL TRIAL: NCT00307996
Title: The Effect of CoQ10 Administration on the Oxidative and Antioxidative Markers in Hemodialysis Patients
Brief Title: The Effect of CoQ10 Administration on Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Shizuoka (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT2006001
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2006-03-28 (Estimated); Status verified 2006-03

CONDITIONS: Chronic Renal Failure; Hemodialysis
Keywords: CoQ10; hemodialysis; oxidative marker; antioxidant
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — coenzyme Q10; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Coenzyme Q10 (drug)

SUMMARY:
The purpose of this study is to examine whether CoQ10 administration is effective as an antioxidant in hemodialysis patients.

DETAILED DESCRIPTION:
Oxidative stress has been recognized as a potential risk factor for such complications as atherosclerosis in hemodialysis patients. This study investigates whether CoQ10 administration is effective for protecting oxidative stress in hemodialysis patients. The subjects were recruited from day-time hemodialysis patients in Iwata City Hospital. 100 mg CoQ10 was administered every HD for 6 months. Several oxidative and antioxidative markers were measured in plasma at pre, 1, 3, 6 months and after washout.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis for at least 6 months

Exclusion Criteria:

* none

Ages: 0 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2004-03; Study Completion 2004-12

PRIMARY OUTCOMES:
Oxidative protein concentration at 6 month
Antioxidant capacity at 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Hiromichi Kumagai, MD, Study Chair — University of Shizuoka
Locations (1):
- Iwata City Hospital, Iwata, Shizuoka, Japan